CLINICAL TRIAL: NCT02434588
Title: Evaluation of an Iris Dilatation Ring in Cataract Surgery
Brief Title: Evaluation of an Iris Dilatation Ring in Cataract Surgery (ADICC-ID)
Acronym: ADICC-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JFO_2014-27; ID-RCB 2014-A01880-47 (Other: ANSM)
Record Dates: First submitted 2015-04-14; First posted 2015-05-05 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Small Pupil
MeSH Terms: conditions — Miosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bhattacharjee ring (Experimental)
  Interventions: Device: Bhattacharjee ring

INTERVENTIONS:
Device: Bhattacharjee ring — Insertion of a Bhattacharjee ring to stabilise the pupil during cataract surgery

SUMMARY:
During cataract surgery, it is necessary to dilate the iris in order to remove the crystalline lens and position the implant. The diameter of the optical implant being 6 mm, in case of capsulorhexis crystalline access 5.5 mm, the expansion should be at least 6 mm.

At pre-operative consultation, the iris is always dilated by instillation of eye drops and measured at the slitlamp. For patients with an inadequate dilation, the intervention requires the use of a mechanical dilatation device.

This study aims to assess the value of an alternative dilatation ring to Malyugin ring, which can be inserted and removed through an incision of less than 2 mm in diameter, due to its size smaller than that of the Malyugin ring.

Our hypothesis is that this Bhattacharjee ring ensures sufficient and stable iris dilation during surgery, enabling implant placement in good conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient with programmed cataract surgery under topical or local anesthesia
* Need to use a dilatation ring during operation, highlighted by iris dilatation ≤ 6 mm on slitlamp, after mydriatic solution and 10% phenylephrine eye drops instillation

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient's refusal to participate in the study
* Patient non covered by health insurance
* Complete iridectomy
* Tearing of iris sphincter
* Important posterior synechiae (when the iris is attached to the anterior surface of the implant)
* Anterior chamber very deep (depth of the anterior chamber lower than 1mm after injection of the viscous product)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with dilated iris ≥ 6 mm | Immediately after ring insertion

SECONDARY OUTCOMES:
Proportion of patients with dilated iris ≥ 6 mm after instillation of dilating eye drops | Immediately before ring insertion
Proportion of patients with ≥ 6mm iris dilation after surgery | Just before ring removal
Proportion of patients with iris retraction ≤ 4 mm immediately | Immediatly after ring removal
Surgeon feeling operational conditions on an visual analogic scale | Immediatly after ring insertion
Change for Malyugin ring during surgery | Just before ring insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rotchschild, Paris, France

REFERENCES:
- [Derived] Salviat F, Febbraro JL, Zuber K, Yavchitz A, Moran S, Gatinel D. Evaluation of a uniplanar pupil expansion ring in small-pupil cataract surgery: a feasibility study. Int Ophthalmol. 2022 Feb;42(2):489-496. doi: 10.1007/s10792-021-02065-9. Epub 2021 Oct 16. PMID 34655377